CLINICAL TRIAL: NCT02496741
Title: Phase Ib Study of Metformin and Chloroquine in IDH1/2-mutated Patients With Glioma, Intrahepatic Cholangiocarcinoma or Chondrosarcoma
Brief Title: Metformin And Chloroquine in IDH1/2-mutated Solid Tumors
Acronym: MACIST
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.W. Wilmink, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBA
Record Dates: First submitted 2015-06-30; First posted 2015-07-14 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Glioma; Cholangiocarcinoma; Chondrosarcoma
Keywords: isocitrate dehydrogenase 1/2 mutation; metformin; chloroquine
MeSH Terms: conditions — Glioma; Cholangiocarcinoma; Chondrosarcoma | interventions — Metformin; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin and chloroquine combination (Experimental): Metformin will be administered in a 3+3 dose-escalation schedule.
  Chloroquine will be administered in a fixed dose.
  Interventions: Drug: Metformin and chloroquine combination

INTERVENTIONS:
Drug: Metformin and chloroquine combination — Metformin and chloroquine are two oral medications. Metformin is to be taken twice daily, chloroquine once daily.
  Other Names: Aralen; Glucophage

SUMMARY:
This phase Ib, open-label, single-center, non-randomized clinical trial will evaluate the toxicity and efficacy of metformin and chloroquine in isocitrate dehydrogenase 1/2-mutated (IDH1/2MT) patients with a glioma, intrahepatic cholangiocarcinoma or chondrosarcoma.

DETAILED DESCRIPTION:
Glioma, intrahepatic cholangiocarcinoma (IHCC) and chondrosarcoma (CS) are aggressive, malignant cancers with a dismal outcome, the two latter types especially in the locally-advanced or metastasized setting. This is due to a lack of effective treatment strategies and highlights the dire need for novel therapies.

A subset of these cancer types are characterized by the presence of mutations in the genes encoding for isocitrate dehydrogenase 1 (IDH1) and isocitrate dehydrogenase 2 (IDH2). These mutations occur in 80% of world health organization (WHO) grade II and III glioma and secondary glioblastoma, 20% of IHCC and 60% of CS and, besides their oncogenic function, induce metabolic vulnerabilities to IDH1/2MT cancer cells that can be exploited in vitro by the oral antidiabetic metformin and the oral antimalarial drug chloroquine.

In the present study protocol, the investigators describe a phase Ib single-center clinical trial in which patients with glioma, IHCC or CS are being screened for IDH1/2MT using the surrogate marker D-2-hydroxyglutarate (D-2HG), which is exclusively produced in IDH1/2MT cancers, or DNA sequencing of tumor material. Eligible IDH1/2MT patients are then treated with a combination of metformin and chloroquine.

The study protocol uses a 3+3 dose-escalation scheme. The primary objective is to determine the maximum tolerated dose in order to establish a recommended dose for a phase II trial. Secondary objectives of the study include (1) to investigate the pharmacokinetics of the combination therapy of metformin plus chloroquine, (2) whether or not IDH1/2MT status can be determined by magnetic resonance spectroscopy and/or mass spectrometry of the serum, urine and/or bile or next-generation sequencing of circulating tumor DNA in glioma, IHCC or CS patients and to (3) investigate the tumor response and D-2HG concentration response to metformin plus chloroquine in IDH1/2MT cancers.

This study may open a novel treatment avenue for IDH1/2MT glioma, IHCC and CS by investigating two relatively safe drugs for these highly malignant tumors. In addition, this study may present novel therapies for other cancers that are regularly affected by IDH1/2MT, such as acute myeloid leukemia, acute lymphocytic leukemia and T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of a glioma, IHCC or WHO grade ≥ II CS (both newly-diagnosed and refractory/relapsed tumors)
2. Tumor carries a neomorphic D-2HG generating mutation in IDH1 or IDH2 as determined by MS of serum and urine (optional: bile), MRS of the tumor or DNA sequencing of (circulating) tumor material.
3. Measurable lesion according to RECIST 1.1 criteria (see Appendix B) in IHCC and CS patients and RANO criteria (see Appendix C) in glioma patients.
4. ECOG/WHO performance 0-2 (see Appendix D).
5. Age > 18 years.
6. Adequate renal function (creatinine < 150 μmol/L and/ or a creatinine clearance > 60 ml/ L).
7. Adequate liver function (bilirubin < 1.5 times upper limit of normal, ALAT or ASAT < 5.0 times upper limit of normal in case of liver metastases and < 2.5 the upper limit of normal in absence of liver metastases).
8. Adequate bone marrow function (WBC > 3.0 x 109/L, platelets > 100 x 109/L).
9. If patient is eligible for resection, surgery is (already) planned at least 4 weeks away from start study treatment.
10. Mentally, physically, and geographically able to undergo treatment and follow up.
11. Signed informed content obtained prior to treatment.

Exclusion Criteria:

1. Pregnancy (positive serum pregnancy test) and lactation.
2. Serious concomitant systemic disorder that would compromise the safety of the patient, at the discretion of the investigator.
3. Patients who have any severe and/or uncontrolled medical conditions such as:

   * unstable angina pectoris,
   * symptomatic congestive heart failure,
   * myocardial infarction,
   * cardiac arrhythmias,
   * pulmonary insufficiency,
   * epilepsy (interaction with chloroquine),
   * severe gastrointestinal, neurological or hematological diseases (interaction with chloroquine).
4. 6 months prior to randomization:

   * serious uncontrolled cardiac arrhythmia,
   * uncontrolled diabetes as defined by fasting serum glucose >2X ULN,
   * active or uncontrolled severe infection, including malaria,
   * cirrhosis, chronic active hepatitis or chronic persistent hepatitis,
   * severely impaired lung function.
5. Patients that use digoxin, MAO inhibitors, fenylbutazone, oxygenbutazone, gold preparations or cimetidine (known pharmaco interaction with chloroquine) or loop diuretics (known pharmaco interaction with metformin) for which no good alternative is available.
6. Patients that have a known history of alcohol abuse (interaction with metformin).
7. Patients with known glucose-6-phosphate dehydrogenase deficiency, porphyria, myasthenia gravis or ocular/retinal aberrations (interaction with chloroquine).
8. Patients with a known hypersensitivity to metformin or chloroquine.
9. Patients that are lactose intolerant.
10. Use of metformin or chloroquine in the previous 6 months.
11. Long-term use of chloroquine (>5 years or cumulative dose >300 grams) in the past.
12. Use of other anti-cancer therapy (i.e. surgical resection, chemotherapy, targeted therapy, radiation therapy, surgery). Palliative therapy is permitted, such as:

    * palliative radiotherapy for symptomatic bone metastases;
    * dexamethasone for symptom relief in patients with glioma and cerebral edema;
    * non-enzyme inducing antiepileptic drugs (with the exception of topiramate) in patients with glioma and epileptic seizures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11; Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of metformin + chloroquine | 1 year
  The maximum tolerated dose is the chloroquine plus metformin dose in which no more than 1 in 3 patients (of a 3+3 dose-escalation schedule) observe serious adverse effects.

SECONDARY OUTCOMES:
Effect of metformin + chloroquine on serum/urine/bile D-2-hydroxyglutarate (D2HG) concentration | 1 year
  D-2HG concentration will be measured by mass spectrometry (MS) in serum/urine/bile, at the beginning and end of the study.
Effect of metformin + chloroquine on intratumoral D2HG concentration | 1 year
  Intratumoral D-2HG concentration will be measured by magnetic resonance spectroscopy (MRS), at the beginning and end of the study.
Effect of metformin + chloroquine on tumor response | 1 year
  Tumor size will be measured using a MRI/CT scan before and after treatment.
Recommended dose of metformin + chloroquine | 1 year
  The recommended dose is the dose of chloroquine plus metformin is the dose level one step below the maximum tolerated dose.

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke W Wilmink, M.D., Ph.D., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (3):
- Netherlands (3):
  - VU University Medical Center, Amsterdam, North Holland
  - Academic Medical Center, Amsterdam, North Holland
  - Leiden University Medical Center, Leiden, South Holland

REFERENCES:
- [Derived] Molenaar RJ, Coelen RJS, Khurshed M, Roos E, Caan MWA, van Linde ME, Kouwenhoven M, Bramer JAM, Bovee JVMG, Mathot RA, Klumpen HJ, van Laarhoven HWM, van Noorden CJF, Vandertop WP, Gelderblom H, van Gulik TM, Wilmink JW. Study protocol of a phase IB/II clinical trial of metformin and chloroquine in patients with IDH1-mutated or IDH2-mutated solid tumours. BMJ Open. 2017 Jun 10;7(6):e014961. doi: 10.1136/bmjopen-2016-014961. PMID 28601826